CLINICAL TRIAL: NCT00302380
Title: An Open Label Phase I/II Study of the Safety and Dopamine Transporter Binding Properties of C-11 Altropane in Normal Human Subjects and in Subjects With ADHD
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Thomas Spencer, MD, Massachusetts General Hospital
Other Study IDs: 2000-p-001975
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A sample of blood (2 tablespoons) will be drawn from all subjects.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- un-medicated subjects with ADHD
  Interventions: Radiation: PET imaging using C-11 altropane as the ligand.
- subjects without ADHD
  Interventions: Radiation: PET imaging using C-11 altropane as the ligand.

INTERVENTIONS:
Radiation: PET imaging using C-11 altropane as the ligand. — A one-injection protocol will be used for the study. C-11 Altropane will be injected manually as an intravenous bolus.

SUMMARY:
The primary objective of this study is to evaluate the Binding Potential in subjects with ADHD and adults without ADHD: the intent being to demonstrate that C-11 Altropane PET can be used to differentiate adults with ADHD from healthy control subjects.

DETAILED DESCRIPTION:
This protocol seeks to replicate and extend our investigation of DAT binding in adults with ADHD with specific aims:

1. To examine dopamine transporter (DAT) receptor binding potential in adults with ADHD, using PET scanning with 11C altropane as the ligand. We hypothesize that compared to adults without ADHD, adults with ADHD will have greater DAT binding that will not be accounted by psychiatric comorbidity or age.
2. To examine the relationship of DAT binding to clinical features of ADHD. We hypothesize that DAT binding will be positively correlated with a) severity of ADHD symptoms and b) neuropsychological and interpersonal dysfunction.
3. To examine the relationship between DAT binding and genetic risk factors. We hypothesize that DAT binding will be specifically associated with homozygosity of the DAT (480) gene in adults with ADHD and not with other ADHD-associated genetic markers (e.g., DRD4-7, D2, DBH).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study.
2. Age: 18 - 55
3. If female, non-pregnant, non-nursing with a negative serum pregnancy test and using an adequate form of birth control.
4. Supine and standing blood pressure within the range 110/60 to 150/90 mmHg.
5. Heart rate, after resting for 5 minutes, within the range 46-90 beats/min.
6. Subjects who are within 20% of the ideal weight for height
7. Right handed
8. Diagnosis of DSM-IV ADHD (current), as manifested in clinical evaluation and confirmed by structured interview (for ADHD study subjects).
9. Subjects without a diagnosis of DSM-IV ADHD (lifetime), as manifested in clinical evaluation and confirmed by structured interview (for control study subjects).

Exclusion Criteria:

1. Diagnosis of any psychotic disorder, bipolar disorder, severe depression, severe anxiety, or Autism. Subjects with mild mood, oppositional, conduct, and anxiety disorders may be permitted to participate if considered appropriate by the investigator
2. Scores of Baseline Scales:

   Hamilton Depression Scale > 17 (out of a possible 67 on the 21-item scale)(Hamilton 1960) Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale)(Beck, Ward et al. 1961) Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale)(Hamilton 1959)
3. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention.
4. Any clinically significant chronic medical condition, in the judgement of the investigator.
5. Mental impairment as evidenced by an I.Q. <75.
6. Subject must be off any investigational drug for at least 4 weeks prior to the start of the study.
7. Exposure to dopamine receptor antagonists, including stimulant medications (e.g. methylphenidate) or buproprion within the previous three (3) months to the start of the study.
8. Exposure to non-stimulant ADHD medications (e.g. atomoxetine) within the previous 4 weeks to the start of the study.
9. Exposure to radiopharmaceuticals within four (4) weeks prior to PET scan.
10. Subjects receiving psychotropic medication.
11. Any clinically significant abnormality in the screening laboratory tests, vital signs, or 12-lead ECG, outside of normal limits.
12. Any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant.
13. Subjects with a known recent history (within the past six (6) months) of illicit drug or alcohol dependence.

Ages: 18 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 200 un-medicated subjects with ADHD and 100 subjects without ADHD will be recruited sequentially. No individual will be excluded based on gender, race, or ethnicity.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2000-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The DAT receptor occupancy of OROS MPH and Metadate CD in adults with and without ADHD using PET scanning with C-11 Altropane. | Subjects will lie still in the PET camera for a 90 minute period.
  PET imaging will be acquired using either a HR+ or Siemens Biograph 64 PET/CT camera.

SECONDARY OUTCOMES:
Neuropsychological tests | Examination of cognitive-neuropsychological functioning will take approximately 2.5 hours to complete.
  Cognitive-neuropsychological functioning will be examined by selected tests that are thought to reflect basic deficits in ADHD, mainly those believed to measure components of attention and prefrontal brain systems.
Genotyping | A sample of blood (2 tablespoons) will be drawn from all subjects.
  Genotyping will be performed using a custom markers for dopamine-related genes (DAT, DRD4-7, D2, and DBH).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Derived] Spencer TJ, Biederman J, Faraone SV, Madras BK, Bonab AA, Dougherty DD, Batchelder H, Clarke A, Fischman AJ. Functional genomics of attention-deficit/hyperactivity disorder (ADHD) risk alleles on dopamine transporter binding in ADHD and healthy control subjects. Biol Psychiatry. 2013 Jul 15;74(2):84-9. doi: 10.1016/j.biopsych.2012.11.010. Epub 2012 Dec 27. PMID 23273726